CLINICAL TRIAL: NCT03829280
Title: Cognitive Adaption Training-Effectiveness in Real-world Settings and Mechanism of Action (CAT-EM)
Acronym: CAT-EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Vanguard Research Group (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dawn Velligan, Henry B. Dielmann Chair of Psychiatry and Behavioral Sciences, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20180237H; 1R01MH117101-01 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Cognitive Adaptation Training; Functional Outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Community Mental Health Services

STUDY DESIGN:
Intervention Model Description: Cluster Randomized clinical trial conducted at 8 community mental health outpatient treatment sites across the country
Who Masked: Outcomes Assessor
Masking Description: Raters assessing clinical outcome variables are centralized raters who are blind to treatment group as well as study design and aims.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Adaptation Training (Experimental): Psychosocial treatment using environmental supports such as signs, alarms, pill containers, checklists, technology and the organization of belongings established in a person's home or work environment to bypass the cognitive and motivational difficulties associated with schizophrenia, and support habits for functional behavior to promote recovery.
  Interventions: Behavioral: Cognitive Adaptation Training
- Community Treatment (Active Comparator): Medication follow-up and case management as provided by the community mental health center according to usual care.
  Interventions: Behavioral: Community Treatment

INTERVENTIONS:
Behavioral: Cognitive Adaptation Training — Psychosocial treatment using environmental supports to bypass cognitive and motivational problems and improve adaptive behavior
  Other Names: CAT
  Arms: Cognitive Adaptation Training
Behavioral: Community Treatment — Medication follow-up and case management as provided in usual community care in the setting
  Other Names: CT
  Arms: Community Treatment

SUMMARY:
The investigators propose a cluster randomized effectiveness trial comparing Cognitive Adaptation Training (CAT; a psychosocial treatment using environmental supports such as signs, alarms, pill containers, checklists, technology and the organization of belongings established in a person's home or work environment to bypass the cognitive and motivational difficulties associated with schizophrenia ) to existing community treatment (CT) for individuals with schizophrenia in 8 community mental health centers across multiple states including 400 participants. Mechanisms of action will be examined. Participants will be assessed at baseline and 6 and 12 months on measures of functional and community outcome, medication adherence, symptoms, habit formation and automaticity, cognition and motivation.

DETAILED DESCRIPTION:
Schizophrenia remains one of the most disabling conditions world-wide with an economic burden that exceeded $155 billion dollars in fiscal year 2013 alone. Despite existing medication and community treatment, many individuals with this diagnosis continue to have poor outcomes and struggle toward recovery. CAT is a psychosocial treatment using environmental supports such as signs, alarms, pill containers, checklists, technology and the organization of belongings established in a person's home or work environment to bypass the cognitive and motivational difficulties associated with schizophrenia, and support habits for functional behavior to promote recovery. In a series of efficacy studies, CAT improved social and occupational functioning, symptoms, and adherence to medication, and reduced rates of readmission. The investigators propose a cluster randomized effectiveness trial comparing Cognitive Adaptation Training (CAT) to existing community treatment (CT) for individuals with schizophrenia in 8 community mental health centers across multiple states including 400 participants. This would be the first large-scale effectiveness study of CAT for improving functional outcomes for those with schizophrenia seen in community mental health centers (CMHCs) where the majority of those with schizophrenia are followed for outpatient care and to study the purported mechanisms of action based on an integrated theoretical model. Participants will be assessed at baseline and 6 and 12 months on measures of functional and community outcome, medication adherence, symptoms, habit formation and automaticity, cognition and motivation. CAT treatment will be weekly for 6 months, biweekly for 3 months and monthly for the remainder of the trial. Purported mechanisms of action for CAT including bypassing impairments in cognitive function to improve functional outcome and bypassing motivational impairments to create automatic habits to improve functional outcome will be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who have given informed consent.
2. Between the ages of 18 and 65.
3. Clinical Diagnosis of Schizophrenia, or Schizoaffective Disorder
4. Able to provide evidence of a stable living environment (individual apartment, family home, board and care facility) within the last three months and no plans to move in the next year.
5. Able to understand and complete rating scales and assessments.
6. Agree to home visits
7. Be able to have reimbursed home visits as part of treatment

Exclusion Criteria:

1. Alcohol or drug or dependence within the past 2 months.
2. Currently being treated by an Assertive Community Treatment (ACT) team.
3. History of assault within the past year or other conditions that in the judgement of the treatment team make home visits unsafe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Social and Occupational Functioning Scale Scores | baseline, 6 months, 12 months
  A rating from 0-100 reflecting global level of Social and Occupational functioning; Higher scores indicate better functioning.

SECONDARY OUTCOMES:
Change in Daily activity | baseline, 6 months, 12 months
  Negative Symptom Assessment item 14 assessing typical daily behavior using a structured interview with behavioral anchor points. Scale is rated 1 to 6 with higher scores indicating lower levels of engagement in daily activity (i.e. more severe apathy)
Change in Multnomah Community Ability Scale mean score | baseline, 6 months, 12 months
  Assessment of community functioning on a 17 -item scale with domains assessing interference with functioning, adjustment to living, social competence and behavioral problems. Items are averaged to produce a mean score. Items are each rated on a scale from 1-5 with higher scores reflecting better community functioning.
Change in Adherence Estimate Score | baseline, 6 months, 12 months
  A 3 item scale assessing variables associated with adherence. Items are rated based upon self report about the importance of taking medication, worry about medication and financial burden of medication on a scale from agree completely to disagree completely. Each answer is assigned points based on an algorithm and added producing a total score. Higher scores indicate a higher risk for adherence and a lower probability of adherence. Scores range for 0 to 100.
Change in Negative Symptom Assessment-16 Mean Score | baseline, 6 months, 12 months
  Assesses 16 negative symptoms in the domains of communication, emotion/affect, social activity, motivation and psychomotor activity on a scale from 1-6. Items are added and divided by 16 to produce a mean score. A global score is also produced based upon clinical judgement following the interview Higher scores reflect higher levels of negative symptoms.
Change in the Expanded Version Brief Psychiatric Rating Scale (BPRS)-total score | baseline, 6 months, 12 months
  24 item scale assessing multiple dimensions of psychopathology including positive symptoms; negative symptoms, anxiety/depression, and activation on a series of 7 point scales. Higher scores reflect higher levels of symptoms.

OTHER OUTCOMES:
Change in Effort Expenditure for Rewards Task (EEfRT) Probability Difference score | baseline, 6 months, 12 months
  computerized task of effort put forth to win various amounts of money under various levels of probability. The probability difference score equals the percent of hard choices in the high probability condition minus the percent of hard choices in the low probability condition. Higher scores indicate more frequent choices of hard tasks at the high versus low probability level. individuals who answer the same way on all tasks are eliminated (estimate 1%)
Change in global score of Brief Assessment of Cognition (BACS) App | baseline, 6 months, 12 months
  Ipad delivered version of BACS assessing memory, attention, executive function and psychomotor speed. Standard scores are generated and summed to create a global cognition score with higher scores indicating better levels of cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Velligan, PhD, Principal Investigator — University of Texas
Locations (8):
- United States (8):
  - United Services Inc., Dayville, Connecticut
  - Henderson Behavioral Health, Lauderdale Lakes, Florida
  - Chestnut Health Systems, Granite City, Illinois
  - Community Mental Health Center Inc., Lawrenceburg, Indiana
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Peace Health, Eugene, Oregon
  - Providence Center, Providence, Rhode Island
  - The Harris Center for Mental Health & IDD, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The investigators will be fully compliant with the NIMH Data Archive Data Sharing Terms and Conditions, including submitting and harmonizing all descriptive/raw data and analyzed data generated by the grant at the item and subject-level to the National Database for Clinical Trials (NDCT). All submitted data will include a Global Unique Identifier (GUID) and will not include personally identifiable information (PII).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 mos following publication of the primary outcomes of the study and extending for a period of 2 years
Access Criteria: deidentified data only upon email request to PI with specific research questions and analysis plan.

DOCUMENTS (1):
  • Informed Consent Form (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03829280/ICF_000.pdf